CLINICAL TRIAL: NCT01971242
Title: A Randomised, Double Blind, Placebo Controlled, Single Centre, 60 Week Trial of Exenatide Once Weekly for the Treatment of Moderate Severity Parkinson's Disease
Brief Title: Trial of Exenatide for Parkinson's Disease
Acronym: EXENATIDE-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013-003363-64
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's; Parkinson's Disease; Exenatide; Bydureon
MeSH Terms: conditions — Parkinson Disease | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide (Active Comparator): Bydureon- 2mg administered subcutaneously once weekly
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): Placebo, 2mg administered subcutaneously once weekly
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Exenatide — 2mg, SC (subcutaneous) once weekly. Number of weeks: 48 weeks. Exenatide is a 39-amino-acid peptide
  Other Names: Bydureon
  Arms: Exenatide
Other: Placebo — Placebo, 2mg, SC (subcutaneous), once weekly for 48 weeks.
  Arms: Placebo

SUMMARY:
This study is a clinical trial in patients with Parkinson's disease, of a drug called Exenatide which is already licensed for the treatment of patients with Type 2 Diabetes. There have been several groups that have confirmed that Exenatide has beneficial effects on nerve cells when tested in the laboratory, that raises the possibility that Exenatide may slow down or stop the degenerative process of Parkinson's disease. In an open label trial in patients with Parkinson's disease who self administered the drug for 1 year, we have previously shown that the drug is well tolerated and shows encouraging effects on the movement and non-movement aspects of the disease, even 2 months after patients stopped administering the drug. The next step is therefore to formally evaluate whether Exenatide really is a potential "neuroprotective" drug, i.e. stops the nerve cells dying in Parkinson's disease, by conducting a double blind, placebo controlled trial.

DETAILED DESCRIPTION:
This trial aims to generate further data to explore whether 48 weeks exposure to Exenatide has an advantage over placebo based on a standard validated assessment of Parkinson's disease severity (the MDS UPDRS part 3 motor subscale). This will be measured during the "practically defined OFF medication state" i.e. after patients have withheld their conventional PD medication overnight. The hypothesis is that Exenatide will be associated with reduced MDS UPDRS part 3 scores at the study end.

To further examine the safety and tolerability of 48 weeks exposure to Exenatide in patients with moderate severity PD.

To collect Pharmacokinetic data regarding the degree of penetration of Exenatide across the blood brain barrier. We hypothesise that any central effects of Exenatide will be mediated through penetration of Exenatide across the blood brain barrier. Data obtained from rodents suggests that blood brain barrier penetration is excellent.

We propose to use a simple parallel group randomised controlled trial design.

No double blind data to support the use of Exenatide are currently available therefore equipoise exists. The null hypothesis is that Exenatide (as Bydureon) has no effect on disease progression.

Initial identification of potential participants- patients attending their routine follow up appointments will be informed about the trial by their neurologist and given a participant information sheet.

Participants who wish to be considered for inclusion in the trial will be screened for eligibility at the National Hospital for Neurology and Neurosurgery, according to inclusion and exclusion criteria. A narrative of what trial participation entails together with the participant information sheet will be used to educate potential participants. Each patient will be aware that they have a 50% chance of being allocated active drug or placebo. They will confirm their willingness to attend the clinic after an overnight period without their conventional PD medication. As part of the informed consent, the contact details of the research team will be given to each patient.

Written informed consent will be obtained from each patient prior to enrollment into the trial. All potential patients will be properly informed as to the purposes of the trial and the potential risks/ benefits known, or that can be reasonably predicted or expected, by an Investigator trained in Good Clinical Practice. The investigator will retain the original copy of the Informed Consent Form signed by the patient, a duplicate will be given to the patient, and a third copy will be filed in the patient's hospital notes. Only the consent form approved by the relevant trial ethics committee will be used.

Randomisation Eligible consenting patients will be randomly allocated into 2 groups to receive either; Bydureon 2mg subcutaneous injection once weekly for 48 weeks n=30, or Bydureon placebo subcutaneous injection once weekly for 48 weeks n=30. Randomisation lists will be sufficiently long to enable continued randomisation should any patients drop out within the first 12 weeks of the study (prior to the first follow up visit).

Withdrawal of medications All patients will continue to have optimal conventional PD medication administered throughout the trial period with the exception of "off medication assessments to be performed at 0,12,24,26,48 and 60 weeks.

Detailed evaluations of all patients will take place at these time points at the National Hospital for Neurology & Neurosurgery (NHNN).

At each assessment the patient will attend the research clinic after an overnight withdrawal from their conventional PD medications to allow an objective measurement of their PD disability. Patients unable to tolerate being off medication will not undergo randomisation.

Blood tests will be performed at each visit. At baseline, Blood tests will include full blood count, urea and electrolytes, liver function tests, thyroid function tests, glucose, HBA1c, amylase and saved serum. At follow up visits, urea and electrolytes, thyroid function, serum amylase will be checked and serum will be stored. These samples are to check both safety and to allow measurement of Exenatide levels to be performed after trial completion.

Urine tests A urine sample will be collected at each visit to allow measurement of exenatide levels after trial completion.

A pregnancy test will also be performed for females of child bearing potential at the baseline visit.

Clinical scales Clinical assessments will be performed at each visit using validated scales to assess movement and non movement aspects of PD. Vital signs and weight will be measured at each visit.

The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS UPDRS).

Part 3 of this scale (motor subscore) will be scored in the absence and presence of conventional PD medication. Part 1,2 & 4 of the scale will also be evaluated in the presence of conventional PD medication (ON state) to evaluate any change in some of the non-motor symptoms of PD, activities of daily living and the complications of chronic PD treatment.

Unified Dyskinesia Rating scale. This is considered to be the most useful and objective way of quantifying dyskinesia severity.

3 day Hauser diary of PD state (Time- On, Off, Troublesome Dyskinesia, Non-troublesome dyskinesia, Asleep). Diary data allows quantification of the amount of time during a 7 day period that patients spend in the varying states of movement ability. Patients will bring with them diaries to quantify their PD control for the preceding 3 days.

Mattis Dementia Rating scale (DRS-2). This scale is a validated global measure of cognitive ability.

Montgomery and Asberg Depression Rating Scale (MADRS). This scale allows for physician quantification of Depression severity.

The PDQ39 (Parkinson's disease questionnaire-39). This is the standard disease specific measure of quality of life in PD comprising 39 questions. It has been extensively validated in previous studies.

Non-Motor Symptoms (NMS) severity scale. This validated scale is a tool to collect data on the frequency and severity of 30 non-motor symptoms sometimes experienced by PD patients.

EQ5D (a standardised instrument for use as a measure of health outcome). This is a simple 5 question form and visual analogue scale that allows calculation of quality adjusted life years (QALY) to enable health economic analyses to be performed

Timed motor tests Patients will be asked to perform a Sit-stand-walk timed test and timed keyboard taps with left and right hand separately, in both the OFF medication and ON medication condition.

The timed Sit-stand-walk test will incorporate time taken from seated position to stand and walk 10 metres, turn and return to original seated position.

Timed keyboard taps will use online website Braintaptest.com to quantify number of alternate taps from key "S" to key ";" using a conventional QWERTY (keyboard layout) keyboard in a 30 second period with each hand in turn. The software is validated and records number of key strokes, dwell time, accuracy & rhythmicity in an automated fashion, is freely available online, allows for coded repeatable assessments which are pseudo-anonymised, and date/time stamped.

Lumbar puncture A lumbar puncture will be performed at 12 weeks and 48 weeks to allow measurement of exenatide levels after trial completion.

DaTSCAN A nuclear medicine scan (DaTSCAN) will be performed at baseline and at the final visit.

Teaching injections Patients will be taught how to self administer injections using online teaching video with support of trained member of the trial team.

Concomitant treatments Trial participants will be permitted to use any licensed PD medication throughout the course of the trial that is recommended by their referring neurologist.

Analyses Adverse events will be reviewed at quarterly trial management group (TMG) meetings and 6 monthly independent Data Monitoring committee (iDMC) meetings. An interim analysis will be performed when the last patient has reached 24 weeks follow up and results presented to the iDMC who will make recommendations to the TMG.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease.
* Males or Females.
* Hoehn and Yahr stage ≤ 2.5 in the On medication state.
* Between 25 and 75 years of age.
* On dopaminergic treatment with wearing off phenomena.
* Ability to self-administer, or to arrange carer administration of trial drug.
* Documented informed consent to participate.

Exclusion Criteria:

* Diagnosis or suspicion of other cause for parkinsonism.
* Body mass index <18.5.
* Known abnormality on CT or MRI brain imaging considered likely to compromise compliance with trial protocol/DaTSCAN acquisition.
* Concurrent dementia defined by a score lower than 120 on the Mattis Dementia Rating Scale.
* Concurrent severe depression defined by a score >16 on the MADRS.
* Prior intra-cerebral surgical intervention for Parkinson's disease.
* Already actively participating in a trial of a device, drug or surgical treatment for Parkinson's disease.
* Severe gastrointestinal disease (e.g. gastroparesis).
* Previous exposure to Exenatide.
* Severely impaired renal function with creatinine clearance <30ml/min.
* History of pancreatitis.
* Hyperlipidaemia.
* History or suspicion of thyroid cancer
* Known or suspected intolerance of DaTSCAN or Potassium Iodide administration.
* Females that are pregnant or breast feeding.
* Participants who lack the capacity to give informed consent
* Any medical or psychiatric condition which in the investigator's opinion compromises the potential participant's ability to participate.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-06; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Efficacy | 60 weeks
  The primary objective is to compare the effectiveness of Exenatide versus placebo on the MDS UPDRS part 3 motor subscale in the "practically defined OFF medication state" in patients with moderate severity PD.

SECONDARY OUTCOMES:
Safety and tolerability | 60 weeks
  • Compare differences at 48 and 60 weeks between the Exenatide and placebo trial arms in:
  * Movement Disorder Society Unified Parkinson's Disease Rating Scale part 1,2,3 and 4 On medication scores
  * Movement Disorder Society Unified Parkinson's Disease Rating Scale part 3 Motor subsection Off medication score at 48 weeks.
  * Mattis Dementia Rating scale (DRS-2).
  * Safety and tolerability of Exenatide as indicated by changes in Vital signs, weight, clinical laboratory measures and Adverse Effects

OTHER OUTCOMES:
Exploratory outcomes | Compare differences at 48 and 60 weeks
  Exploratory outcomes:
  • Compare differences at 48 and 60 weeks between the Exenatide and placebo trial arms in:
  * Unified Dyskinesia Rating scale
  * 3 day Hauser diary of PD state (Time-On, Off, Non troublesome Dyskinesia, Troublesome dyskinesia, Asleep)
  * Montgomery and Asberg Depression Rating Scale (MADRS)
  * Parkinson's Disease 39 item Quality of life questionnaire (PDQ39)
  * Non-Motor Symptoms scale (NMSS)
  * Levodopa equivalent doses (LED)
  * Quantitative change in Dopamine Transporter availability as measured by DaTSCAN uptake between baseline and 60 week evaluations
  * Exenatide level in blood, urine every 12 weeks, CSF (at 12 and 48 weeks)
  * CSF levels of BDNF (at 12 and 48 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Foltynie, Dr, Principal Investigator — UCL Institute of Neurology
Locations (1):
- National Hospital for Neurology & Neurosurgery (part of UCLH NHS Trust), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share individual participant data (IPD)

REFERENCES:
- [Derived] Athauda D, Maclagan K, Skene SS, Bajwa-Joseph M, Letchford D, Chowdhury K, Hibbert S, Budnik N, Zampedri L, Dickson J, Li Y, Aviles-Olmos I, Warner TT, Limousin P, Lees AJ, Greig NH, Tebbs S, Foltynie T. Exenatide once weekly versus placebo in Parkinson's disease: a randomised, double-blind, placebo-controlled trial. Lancet. 2017 Oct 7;390(10103):1664-1675. doi: 10.1016/S0140-6736(17)31585-4. Epub 2017 Aug 3. PMID 28781108